CLINICAL TRIAL: NCT01456598
Title: Prospective Multicenter Randomized Controlled Clinical Trial for Comparison Between Laparoscopic and Open Subtotal Gastrectomy With D2 Lymph Node Dissection for Locally Advanced Gastric Cancer
Brief Title: Efficacy of Laparoscopic Subtotal Gastrectomy With D2 Lymph Node Dissection for Locally Advanced Gastric Cancer
Acronym: KLASS-02-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Sang-Uk Han, Professor, Department of Surgery, Ajou University School of Medicine, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-MED-MDB-11-233
Record Dates: First submitted 2011-10-11; First posted 2011-10-21 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Gastric Cancer
Keywords: Stomach neoplasm; Laparoscopy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic gastrectomy (Experimental): Laparoscopic subtotal gastrectomy and D2 lymph node dissection are performed for locally advanced gastric cancer.
  Interventions: Procedure: Laparoscopic gastrectomy
- Open gastrectomy (Active Comparator): Open subtotal gastrectomy and D2 lymph node dissection are performed for locally advanced gastric cancer.
  Interventions: Procedure: Open gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic gastrectomy — * After laparoscopic observation, the possibility of surgery can be considered by examining inside of abdomen.
  * The surgeon undergoes laparoscopic subtotal gastrectomy and D2 lymph node dissection
  * After lymph node dissection, it is possible to undergo gastrectomy on appropriate part and reconstruction under small incision or laparoscopic view.
  * As the reconstruction, one of the techniques like Billroth I, Billroth II and Roux en Y and so on is applied and there is no limitation on use of appliance.
  Other Names: Group A; LDG
  Arms: Laparoscopic gastrectomy
Procedure: Open gastrectomy — * After laparotomy, the possibility of surgery can be considered by examining inside of abdomen.
  * The surgeon undergoes open subtotal gastrectomy and D2 lymph node dissection
  * After lymph node dissection, one of the techniques likes Billroth I, Billroth II and Roux en Y and so on is applied and there is no limitation on use of appliance.
  Other Names: Group B; ODG
  Arms: Open gastrectomy

SUMMARY:
* It was confirmed that the laparoscopic surgery decreases the postoperative pain and reduces the recovery periods in the various surgical fields such as cholecystectomy and colectomy etc. Also, there are clinical evidences that the laparoscopic surgery is applicable to malignant tumor according to the development of surgical techniques and medical instruments.
* In case of early stage of gastric cancer, as the diverse clinical evidences, the gastrectomy has been commonly applied, however, the opening surgery is still applied for advanced gastric cancer due to lack of clinical evidence.
* In Korea, approximately 38% of patients who undergo surgery for gastric cancer are diagnosed by T2-T3 (AJCC 6th edition) (www.i-kgca.or.kr, National gastric cancer registration business in 2009). There are various clinical evidences to apply laparoscopic surgery to the patients, however, most of them are retrospective or cohort study results.
* For the clinical application of surgical treatment regarding locally advanced gastric cancer using laparoscopic surgical technique, it requires the confirmation of definite execution for laparoscopic gastrectomy and D2 lymph node dissection and the safety of surgery and oncological usefulness should be verified.
* In order for this, it is only possible to confirm through the comparison of short-term surgical results (complications, mortalities, operative time and duration of hospitalization etc) and long-term results (survival rates and recurrence rates etc) between laparoscopic surgery and opening surgery based on the multicenter large-sized randomized prospective study with current standard treatment.

DETAILED DESCRIPTION:
Participating Surgeons

* Prior to this clinical trial, only the surgeons who are considered to have the standardization by participating the assignment entitled with "KLASS-02-QC: Standardization of D2 Lymphadenectomy and Surgical Quality Control for KLASS-02 Trial"(ClinicalTrials.gov No: NCT01283893).

Patients Registration

* It is required to ensure that the patients meet the inclusion criteria for this clinical trial, are free from any items of exclusion criteria, are explained about the participation in the clinical trial along with the informed consent forms.
* After rechecking the patients with the registration check list by accessing the web-based randomized program provided from Ajou University clinical trial center.

Randomization

* The registration randomization should be done with 1:1 ratio for each researcher.
* Baseline number (BN) should be provided to the subjects in the order of acquisition of informed consent form. Based on the subjects who are selected as the appropriate subjects in the end, the allocation number (AN) shall be provided in the order of randomized allocation table.

Procedure

* Operations are performed according to the allocated group.

Adjuvant Treatment

* If it is under Stage II and Stage III in the final postoperative pathology, the adjuvant chemotherapy based on 5-FU.

Evaluation of efficacy and safety

* 3-year Relapse free survival rate and overall survival rate of the patients who undergo laparoscopic and open subtotal gastrectomy and D2 lymph node dissection.
* Analysis of recovery after laparoscopic and open subtotal gastrectomy and D2 lymph node dissection.
* Postoperative complications of the patients who undergo laparoscopic and open subtotal gastrectomy and D2 lymph node dissection within postoperative 3 weeks and later.
* The quality of life at preoperative, postoperative 25 days and 1 years using recovery index such as recovery of postoperative intestinal hypermotility, meals and duration of hospitalization, EORTC-C30 and STO22 questionnaire between the patients who underwent laparoscopic and open subtotal gastrectomy and D2 lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* The patient from over 20 years to under 80 years
* The patient with the capability for ECOG (Eastern Cooperative Oncology Group performance status) is ranged between 0 and 1
* The patient included between ASA score (American society of anesthesiology) class I and III
* The patient who is diagnosed as gastric adenocarcinoma under preoperative endoscopic biopsy
* The patient who is diagnosed as locally advanced gastric cancer with the suspicious infiltration of over muscular layer without infiltration on adjacent organs, and without or with lymph node metastasis limited to perigastric or around stomach left gastric artery at the preoperative examination.
* The patient who is suitable for subtotal resection in the preoperative examination
* The patient who is fully explained about purpose of trial and contents prior to the participation into this study and signed on the informed consent approved by Institutional Review Board according to own opinion

Exclusion Criteria:

* The patient who shows distant metastasis under preoperative examination
* The patient with medical history for gastrectomy in the past
* The patient with complication (complete obstruction and perforation) by gastric cancer
* The patient who undergoes anticancer or radiologic therapy prior to the operation or who undergoes endoscopic submucous dissection for currently diagnosed gastric cancer
* The patient who undergoes surgery or anti-cancer radiologic therapy for primary cancer within 5 years
* Vulnerable patients (lack of capacity for decision making, pregnant women (or under planning))
* The patient who has participated into another clinical trial within recent 6 months or who is participating into another trial
* The patient with double cancer of activity and synchronization

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2011-11-21 (Actual); Primary Completion 2018-06-02 (Actual); Study Completion 2018-06-02 (Actual)

PRIMARY OUTCOMES:
3 year relapse free survival | 36 months
  In terms of locally advanced gastric cancer, to examine the non-inferiority of disease free sur-vival rate in laparoscopic subtotal gastrectomy with D2 lymph node dissection at postoperative 3 years compared with open subtotal gastrectomy with D2 lymph node dissection

SECONDARY OUTCOMES:
Early postoperative complication | 3 weeks
  Early postoperative complication is defined as the events which occurs with-in postoperative 21 days, extension of hospitalization and rehospitaliation. It is necessary to evaluate the complication and if it occurs during the hospitalization, it is required to record complication name and date of on-set (postoperatively) and treatment for complication.
Postoperative mortality | 90 days
  It is defined as the death within postoperative 90 days regardless of postoperative reason. If the patient is transferred to other medication institutes with impossible condition for revocery be-fore death, it is regarded as death.
Late postoperative complication | 36 months
  Late postoperative complication is defined the events which occurs after postoperative 21 days. It is necessary to evaluate the complication. it is required to record complication name and date of on-set (postoperatively) and treatment for complication.
Postoperative recovery index | 4 weeks
  Postoperatively, the examiner evaluates the patient's recovery condition (gas exhaust) once a day. Evaluation items for patient's recovery condition: record the meal process once a day and inquire the pain score (10-scored scale) and blood test results during postoperative hospitalization.
Postoperative quality of life | preoperative, 3 weeks, 12 months
  On preoperative, postoperative 3 weeks and postoperative 12 months, both EORTC-C30 and STO22 are analyzed with quality of life by following methods. In case of EORTC-C30, the analysis is undergone by classifying into 5 functional scales (physical, role, emotional, cognitive, and social fungtioning), 3 symptom scales (fatigue, pain and nausea, and vomiting), 1 global health status and 6 single items.
3 years overall survival | 6, 12, 18, 24, 30 and 36 months
  As one of the secondary endpoints, the overall survival rate in laparoscopic subtotal gastrectomy with D2 lymph node dissection at postoperative 3 years compared with open subtotal gastrectomy with D2 lymph node dissection. The schedule of visit is based on every 3 months for 3 years. If subjects cannot visit every 3 months, the investigator can arrange the schedule. However, enrolled should visit every 6 months for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: San-Uk Han, M.D., Ph.D., Principal Investigator — Department of Surgery, Ajou University School of Medicine
Locations (13):
- South Korea (13):
  - Department of Surgery , SOON CHUN HYANG UNIVESITY HOSPITAL, Bucheon-si
  - Keimyung University Dongsan Medical Center, Daegu
  - Copyright National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - Incheon St, Mary's Hostpial, The Catholic University of Korea, Incheon
  - Dong-A University Hospital, Pusan
  - Department of Surgery, Seoul National University BUNDANG Hospital, Seongnam
  - Department of Surgery, Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Yeoeuido St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Department of surgery, GANGNAM SEVERANCE HOSPITAL, Seoul
  - EWHA Womans university medical center, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Background] Kim W, Song KY, Lee HJ, Han SU, Hyung WJ, Cho GS. The impact of comorbidity on surgical outcomes in laparoscopy-assisted distal gastrectomy: a retrospective analysis of multicenter results. Ann Surg. 2008 Nov;248(5):793-9. doi: 10.1097/SLA.0b013e3181887516. PMID 18948806
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Derived] Son SY, Hur H, Hyung WJ, Park YK, Lee HJ, An JY, Kim W, Kim HI, Kim HH, Ryu SW, Kim MC, Kong SH, Cho GS, Kim JJ, Park DJ, Ryu KW, Kim YW, Kim JW, Lee JH, Yang HK, Han SU; Korean Laparoendoscopic Gastrointestinal Surgery Study (KLASS) Group. Laparoscopic vs Open Distal Gastrectomy for Locally Advanced Gastric Cancer: 5-Year Outcomes of the KLASS-02 Randomized Clinical Trial. JAMA Surg. 2022 Oct 1;157(10):879-886. doi: 10.1001/jamasurg.2022.2749. PMID 35857305
- [Derived] Hyung WJ, Yang HK, Park YK, Lee HJ, An JY, Kim W, Kim HI, Kim HH, Ryu SW, Hur H, Kim MC, Kong SH, Cho GS, Kim JJ, Park DJ, Ryu KW, Kim YW, Kim JW, Lee JH, Han SU; Korean Laparoendoscopic Gastrointestinal Surgery Study Group. Long-Term Outcomes of Laparoscopic Distal Gastrectomy for Locally Advanced Gastric Cancer: The KLASS-02-RCT Randomized Clinical Trial. J Clin Oncol. 2020 Oct 1;38(28):3304-3313. doi: 10.1200/JCO.20.01210. Epub 2020 Aug 20. PMID 32816629
- See also: Institutional Review Board, Ajou University Hospital — https://eirb.ajoumc.or.kr/
- See also: The Korean Gastric Cancer Association — http://www.kgca-i.or.kr/html/